CLINICAL TRIAL: NCT02276911
Title: Safety and Efficacy of Pre-incisional Intravenous Ibuprofen to Reduce Postoperative Pain and Opioid Dependence After Posterior Cervical or Lumbar Instrumented Spine Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No enrollment
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Principal Investigator, Lori Wood, Clinical Research Operations Manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13BN033
Record Dates: First submitted 2014-10-22; First posted 2014-10-28 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cervical Spondylosis; Lumbar Spondylosis
MeSH Terms: conditions — Spondylosis | interventions — Ibuprofen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous (IV) ibuprofen (Active Comparator): 800mg IV ibuprofen before incision, followed by four total scheduled doses of IV ibuprofen every six hours for 24 hours, in addition to whatever narcotic or other pain control regimens prescribed by the treating physician to control postoperative pain.
  Interventions: Drug: Ibuprofen
- Intravenous (IV) normal saline (Placebo Comparator): 800mg normal saline before incision, followed by four total scheduled doses of IV ibuprofen every six hours for 24 hours, in addition to whatever narcotic or other pain control regimens prescribed by the treating physician to control postoperative pain.
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Ibuprofen
  Other Names: Caldolor
  Arms: Intravenous (IV) ibuprofen
Other: normal saline
  Other Names: NS
  Arms: Intravenous (IV) normal saline

SUMMARY:
A prospective, randomized, placebo controlled, double-blinded study at a single institution.

DETAILED DESCRIPTION:
Pain medicine literature and the principal investigator's anecdotal experience in posterior cervical and lumbar instrumented spine surgery suggest that pre-incisional IV ibuprofen significantly reduces postoperative pain without increasing surgical complications or fusion rate, which leads to earlier ambulation, less dependence on narcotic medications, shorter hospital stays, and earlier return to work. The purpose of this study is to assess if these anecdotal findings hold true in a randomized clinical trial of patients with cervical or lumbar spondylosis, who are undergoing decompression and instrumented fusion of the spine.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Able to give consent
* Diagnosed with spondylosis, stenosis, and/or instability of the cervical spine
* Diagnosed with spondylosis, stenosis, and/or instability of the lumbar spine
* Require a posterior decompression with internal fixation
* Likely to complete the trial

Exclusion Criteria:

* Patients with previous surgery at the treated spine segment
* Women who are pregnant or plan to become pregnant during the study period Renal/liver disease
* Anemia; coagulopathy
* Thrombocytopenia (<30,000)
* Coronary artery disease
* Previous coronary artery bypass graft (CABG)
* Patients taking Coumadin, Plavix, Lithium, or ACE-inhibitors plus Lasix; non-steroidal anti-inflammatory drug (NSAID) hypersensitivity
* Gastric ulcers
* Recent stroke
* Traumatic brain injury, or intracranial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Change in pain level | pre-operative, 1-3 weeks post-operative, 6 months post-operative
  Visual Analog Scale (VAS) scores at rest and with movement, Macqill Pain Questionnaire scores, and total morphine and morphine equivalents used during hospital admission.
Change in overall health/function | pre-operative, 1-3 weeks post-operative, 6 months post-operative
  SF-36 scores, total length of hospital stay, time to ambulation, and time to return to work.
Fusion rates | 6 month post-operative
  Assessed by plain x-rays or CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Theodore, MD, Principal Investigator — St. Joseph Hospital and Medical Center
Locations (1):
- SJHMC/Barrow Neurosurgical Associates, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
The study was closed due to low enrollment. There was no data analysis done so there will be no information to share.